CLINICAL TRIAL: NCT04034446
Title: a Feasibility and Safety Study of Bispecific CD19-CD22 CAR-T Cell in the Treatment of Relapsed or Refractory B-ALL
Brief Title: CD19-CD22 Chimeric Antigen Receptor T (CAR-T) Cell for Treatment of B Cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to adjustments in the company's strategy, the research and development of this project has been terminated.
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT2019005
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2020-05

CONDITIONS: Relapsed or Refractory B Cell Acute Lymphoblastic Leukemia
Keywords: Relapsed; Refractory; B-ALL
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A (Experimental): Single dose of CD19-CD22 CAR-T cells
  Interventions: Biological: CD19-CD22 CAR-T cells

INTERVENTIONS:
Biological: CD19-CD22 CAR-T cells — 0.5 to 3.0 x 106 autologous CD19-CD22 CAR-T cells per kg body weight, with a maximum dose of 4 x 108 autologous CD19-CD22 CAR-T cells via intravenous infusion.

SUMMARY:
This is a single arm, open-label, single center study to determine the safety and efficacy of CD19-CD22 CAR-T cells in patients with CD19+CD22+ Leukemia.

DETAILED DESCRIPTION:
This is a single arm, open-label, single center study to determine the safety and efficacy of CD19-CD22 CAR-T cells in patients with relapsed or refractory B-ALL. The study will have the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up, and Survival Follow-up. The total duration of the study is 2 years from CD19-CD22 CAR-T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is signed by a subject or his lineal relation.
2. Age 3 and older.
3. Documentation of cluster of differentiation 19 (CD19) and or cluster of differentiation 19 (CD22) expression on leukemic blasts in the BM, peripheral blood within 3 months of screening.;
4. Relapsed or refractory B-cell ALL

   * Relapse within 12 months of first remission
   * Without remission after 2 cycles of induction chemotherapy regimen.
   * Without remission or relapse after salvage treatments.
   * Any BM relapse after autologous stem cell transplantation (ASCT).
5. Without remission or relapse after any prior CD19 targeted therapy;
6. Patients with Philadelphia chromosome positive (Ph+) ALL are eligible if they are intolerant to or have failed 2 lines of tyrosine kinase inhibitor therapy (TKI); no TKI salvage treatments if the patient has a BCR-ABL1 kinase domain gatekeeper mutation Thr315Ile (T315I) mutation.
7. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening；
8. Eastern cooperative oncology group (ECOG) performance status of 0 to 2.
9. Adequate organ function defined as:

   * Aspartate aminotransferase (AST) ≤3 upper limit of normal (ULN);
   * Serum alanine aminotransferase (ALT) ≤3 ULN;
   * Total bilirubin ≤ 2 ULN, except in individuals with Gilbert's syndrome;
   * Note: Patients with Gilbert's syndrome that bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN will be eligible.
   * A serum creatinine≤ 1.5 ULN or Creatine removal rate ≥ 60mL/min（Cockcroft and Gault）
   * Must have a minimum level of pulmonary reserve as ≤ Grade 1 dyspnea and oxygen saturation > 91% on room air.
   * Absolute lymphocyte count ≥0.3 x 10⁹/L.
10. Women of child-bearing potential and all male participants must use highly effective methods of contraception for a period of 1 year after the CD19-CD22 CAR-T cells infusion.

Exclusion Criteria:

1. Active central nervous system leukemia
2. Patients with evidence of currently uncontrollable serious active infections (e.g., sepsis, bacteremia, fungemia, viremia, etc.).
3. Patients who are positive for any of HIV antibody, TP antibody, hepatitis B surface antigen (HBsAg) and hepatitis C virus (HCV) antibody.
4. Major surgery within ≤ 4 weeks before enrollment.
5. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent.
6. Impaired cardiac function:

   * Left Ventricular Ejection Fraction (LVEF) ≤45%;
   * III/IV congestive heart failure (NYHA);
   * Severe arrhythmia (except for Atrial fibrillation, Paroxysmal supraventricular tachycardia);
   * Corrected QT interval (QTc) ≥450ms (male) or QTc≥470ms (female)（QTc using Bazett's formula (QTcB)=QT/RR^0.5）;
   * Myocardial infarction or Coronary Artery Bypass Graft Surgery, heart stent surgery.
   * Other heart diseases that have been judged by the investigator to be unsuitable for receiving cell therapy.
7. Patients with a history of epilepsy or other active central nervous system diseases.
8. Life expectancy < 12 weeks.
9. Allergy to macromolecule biopharmaceuticals such as antibodies or cytokines.
10. Subjects who are receiving systemic steroid treatment and who have been determined by the researchers to require long-term treatment with systemic steroids during treatment, and subjects treated with systemic steroids must be excluded < 72 hours prior to CNCT19 infusion (except inhalation or local use).
11. Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months
Overall remission rate (ORR) | 3 months

SECONDARY OUTCOMES:
Response at Day 28 days | 1 month
Percentage of patients who achieve complete remission (CR) or complete remission with incomplete blood count recovery (CRi) at month 6 without SCT between CD19-CD22 CAR-T cells infusion and Month 6 response assessment. | 6 months
Percentage of patients who achieve CR or CRi with minimal residual disease (MRD) negative bone marrow | 6 months
Relapse-free survival (RFS) | 24 months
Duration of remission (DOR) | 24 months
Overall survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China